CLINICAL TRIAL: NCT00476502
Title: Study of Genetic Polymorphisms of CYP 3A and MDR-1 Genes in Thai HIV-1 Infected Patients on Saquinavir/Ritonavir
Brief Title: Study of Genetic Polymorphisms in Thai HIV-1 Infected Patients on SQV/r
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 031
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
Keywords: genetic polymorphism; CYP 3A; MDR-1; Thai; HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — PBMC
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: patients involved in structured interruption therapy
  Interventions: Genetic: identify genetic polymorphism in Thai HIV infected

INTERVENTIONS:
Genetic: identify genetic polymorphism in Thai HIV infected — Gene sequencing of Cyp450 metabolic pathway

SUMMARY:
Study of genetic polymorphisms of CYP #A and MDR-1 genes in Thai HIV-1 infected patients on saquinavir/ritonavir.

DETAILED DESCRIPTION:
Genetic polymorphisms will be investigated by polymerase-chain reaction (PCR) and drug levels of saquinavir will be determined by high phase liquid chromatography with UV-detected (HPLC).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected persons who have been enrolled in the Staccato study
* On low-dose ritonavir boosted saquinavir at the time blood samples are collected

Exclusion Criteria:

* Inability to understand the nature and extent of the study and the procedures required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients on stable SQV based HAART therapy
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)
Locations (1):
- The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok, Bangkok, Thailand

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org